CLINICAL TRIAL: NCT05855720
Title: Bundesweit Einheitliche Wissenschaftliche Evaluation Von Modellvorhaben Nach § 64b SGB V ab 2022
Brief Title: Nationwide Uniform Scientific Evaluation of Flexible and Integrated Treatment Projects From 2022 Onwards
Acronym: EVA64_2
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: Institute of Social Medicine and Health Services Research, Medical Faculty, Otto-von-Guericke- University Magdeburg, Germany (Unknown); WIG2 Scientific Institute for Health Economics and Health System Research Leipzig, Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: EVA64.2
Record Dates: First submitted 2023-05-04; First posted 2023-05-11 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Mental Health; Cross-sectoral Treatment; Flexible and Integrated Treatment; FIT; Psychiatry; Evaluation Study; Cohort Studies
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group (IG): Patients being treated in FIT model project
  Interventions: Other: FIT model project
- Control Group (CG): Patients being treated in standard care (control hospitals)

INTERVENTIONS:
Other: FIT model project — Several statutory health insurance (SHI) funds have established contracts with hospitals for an alternative remuneration / financing of patients treated in the hospital (FIT hospital). Some of those contracts already started in 2013 and were prolonged. Some FIT contracts will start freshly (until June 2026). These contracts encourage FIT hospitals to test alternative treatment options for their patients (insured with the involved SHI funds), for example fewer inpatient and more outpatient treatment.
  Groups: Intervention Group (IG)

SUMMARY:
This study is an evaluation of flexible and integrated psychiatric care models (according to § 64b of the German Social Code Book V (SGB V)) (FIT) including new FIT projects starting after 2022 and the prolongation of any of 19 already established FIT projects (mainly at German psychiatric hospitals). The central concern of this evaluation is to answer the question whether FIT care offers advantages over standard care. The orientation of model care is a more cross-sectoral provision of services through more flexible psychiatric treatment intensities. However, FIT program structures depend on the individual situation and organization of the FIT hospital together with the participating statutory health insurance (SHI) funds.

DETAILED DESCRIPTION:
The introduction of Section 64b of the German Social Code, Book V (SGB V) created the possibility of agreeing so-called FIT (flexible and integrated treatment) model projects for the further development of care for mentally ill people in Germany. The objective is to improve cross-sectoral care or optimize patient care. More than 20 FIT projects have been established at German psychiatric hospitals since 2013. Some FIT projects were prolonged after eight years (max. 15 years in sum). New FIT projects are planned.

In accordance with § 65 SGB V, all FIT projects under § 64b SGB V, must be scientifically evaluated by an independent expert. The aim of this evaluation is to examine the achievement of the objectives of the FIT model projects based on anonymized claims data.

The effectiveness, costs, and cost-effectiveness of the FIT model hospital care compared to standard care are to be examined. FIT projects include those starting before 2022 and being prolonged and those FIT projects starting between 2022 and June 2026. The study presented here is a controlled cohort study utilizing anonymous claims data. The controlled design is based on the fact that information of patients from intervention hospitals (any FIT design) is compared to information of comparable patients from structurally similar psychiatric hospitals in the same federal state (Petzold et al, Gesundheitswesen 2019, 81(1):63-71).

ELIGIBILITY:
Inclusion Criteria:

* treatment in any of the participating hospitals or control hospitals within recruitment phase (number of hospitals will be fix until June 2026)
* being insured with any of the participating SHI funds

Exclusion Criteria:

* less than one year follow-up data available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: anonymized data of the participating SHI funds, all patients being treated in any of the participating FIT hospitals (within FIT model period) or a control hospital within recruitment period
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2038-12 (Estimated); Study Completion 2041-07 (Estimated)

PRIMARY OUTCOMES:
Duration of inpatient psychiatric treatment | one year prior to recruitment compared to first to max year after recruitment. Max year = latest possible year for maximal observation period depending on the length of FIT project
  Days with inpatient stays of each included patient will be marked within the patient-individual follow-up period. A billing matrix defining the type of charge and describing the count will be used to mark days with inpatient stays. Inpatient stays that range outside the patient-specific follow-up time will be censored. The proportion of patients with at least one inpatient stay will be presented. Furthermore, the days of inpatient stays per patient will be added, including the stay that led to inclusion in the evaluation. The classification into inpatient and day care is based on the corresponding charges. If inpatient and day care cases are billed on one day in one hospital, this day will be counted as an inpatient day. It will be analyzed how long patients were treated in hospitals (here only inpatient stays), summed over the entire observation period for each case (all patients).
Sick leave days | one year prior to recruitment compared to first to fourth year after recruitment
  The number of sick leave days due to any mental disorder will be counted.

SECONDARY OUTCOMES:
Duration of day care psychiatric treatment | one year prior to recruitment compared to first to max year after recruitment
  Days with day care stays of each included patient will be marked within the patient-individual follow-up period. A billing matrix defining the type of charge and describing the count will be used to mark days with day care stays. Day care stays that range outside the patient-specific follow-up time will be censored. The proportion of patients with at least one day care stay will be presented. Furthermore, the days of day care stays per patient will be added, including the stay that led to inclusion in the evaluation. The classification into inpatient and day care is based on the corresponding charges. If inpatient and day care cases are billed on one day in one hospital, this day will be counted as an inpatient day. It will be analyzed how long patients were treated in hospitals (here only day care stays), summed over the entire observation period for each case (all patients).
Outpatient psychiatric treatment (within and outside the hospital) | one year prior to recruitment compared to first to max year after recruitment
  The number of days with a contact in the psychiatric outpatients departments (PIA) and with outpatient treatment due to any psychiatric treatment of patients treated in the IG and CG will be recorded and compared.
Continuity of care | one year prior to recruitment compared to first to max year after recruitment
  It will be analyzed how many cases had at least one contact with the outpatient sector after hospital discharge. A distinction will be made between the outpatient sector in the hospital (PIA) and the outpatient sector outside the hospital (contracted medical sector). In addition, the area of continuity of treatment in the "psychiatric sector" (PIA, physician for psychiatry or child and adolescent psychiatry or psychotherapist) will be summarized.
Inpatient hospital readmission | one year prior to one year after first full inpatient psychiatric discharge after recruitment
  The proportion of persons with an inpatient stay who were readmitted as inpatients within one year after discharge from the hospital and the days between first inpatient discharge and second inpatient treatment will be examined. The follow-up period is determined on a patient-specific basis. For this purpose, the first discharge date from an inpatient stay in the reference hospital (IG or CG) after inclusion into the evaluation that allowed a one-year follow-up period will be taken as the basis. Readmission is given if the patient had a hospital stay with any psychiatric diagnosis as main diagnosis and was readmitted with a psychiatric diagnosis as main diagnosis within one year.
Discontinuation of contacts for severely mentally ill patients within the psychiatric care system | one year prior to one year after recruitment
  The frequency of severely mentally ill patients with no contact to the psychiatric care system within 90 and 180 days will be investigated.
Hopping | one year prior to recruitment compared to first to max year after recruitment
  The percentage of patients with more than three different service providers within the same care sector will be investigated.
Comorbidities | one year prior to recruitment compared to first to max year after recruitment
  The number of comorbidities will be determined for each patient within the follow-up period and compared between IG and CG. Comorbidities are defined based on the diagnoses of the Elixhauser Score, the diagnosis groups are added unweighted in the context of this analysis.
Mortality | event time analysis
  The proportion of individuals who die within a defined period of time after inclusion in the evaluation will be analyzed.
Disease progression | event time analysis
  The proportion of patients who transition from F32.0 or F32.1 (mild/moderate depressive episode) to F32.2 or F32.3 (severe depressive episode) or from F32 (depressive episode) to F33 (recurrent depressive disorder) or from no addictive disorder (F10-F19) to any additive disorder (F10-F19) will be recorded.
Direct medical care costs | one year prior to recruitment compared to first to max year after recruitment
  The difference in the costs for the treatment of mental illnesses arising between IG and CG during the observation period will be analyzed. In addition, somatic costs will be estimated. For this purpose, the care costs of the following areas will be taken into account: costs of inpatient and day care, cost of outpatient care in hospitals, costs of SHI-accredited medical care, drug costs and remedies costs.
Cost-effectiveness (direct medical costs) | one year prior to recruitment compared to first to max year after recruitment
  To compare the efficiency of the model project with standard care, a cost-effectiveness analysis will be performed taking a SHI-funds perspective. The incremental cost-effectiveness ratio will be determined using the primary outcome parameter cumulative duration of inpatient stays as the effect measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Social Medicine and Health System Research (ISMG), Medical Faculty, Otto-von-Guericke-University Magdeburg, Magdeburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petzold T, Neumann A, Seifert M, Kuster D, Pfennig A, Weiss J, Hackl D, Swart E, Schmitt J. [Identification of Control Hospitals for the Implementation of the Nationwide and Standardized Evaluation of Model Projects According to section sign 64b SGB V: Analysis of Data from Structured Quality Reports]. Gesundheitswesen. 2019 Jan;81(1):63-71. doi: 10.1055/s-0042-116436. Epub 2016 Nov 15. German. PMID 27846670